CLINICAL TRIAL: NCT05431660
Title: Effects of Diabetic Foot School on Sensory, Balance and Lower Extremity Biomechanics
Brief Title: Diabetic Foot School and Biomechanics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-587/35
Record Dates: First submitted 2022-05-25; First posted 2022-06-24 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Educational Status; Control Groups

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: The people participating in the study will not know in which group they are in the study, but since the physiotherapist who gives the training and gives the treatment is the only person, the study will continue as a single blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tele-rehabilitation group (Experimental): 1st group within the scope of diabetic foot school, and an exercise program aiming to increase the mobility and strength of the foot will be implemented through video calls twice a week, face-to-face once a week for 8 weeks.
  Interventions: Other: education and exercise protocol about diabetic foot
- face to face training group (Active Comparator): The 2nd group will be given a booklet covering this training and they will be followed up with video calls 1 day a week for 8 weeks.
  Interventions: Other: control group

INTERVENTIONS:
Other: education and exercise protocol about diabetic foot — In diabetic foot school education, foot anatomy and functions, biomechanics, diabetic foot causes, epidemiology, causes of pain will be explained and treatment methods, ergonomic information, exercises to be done, sensory education, appropriate positions in daily life activities, risky situations, points to be considered and foot care. information will be given.
  Arms: tele-rehabilitation group
Other: control group — diabetic foot school information booklet and weekly video conference meeting
  Arms: face to face training group

SUMMARY:
The primary aim of the study is to establish a diabetic foot school. The secondary aim is to compare the effects of the training given to diabetic foot patients within the scope of the diabetic foot school, on sensory, balance, lower extremity biomechanics and the effectiveness of these individuals on the knowledge level of diabetic foot.

With the evaluations to be made, the effectiveness of the diabetic foot school program will be proven and it will contribute to the literature with objective and evidence-based results. For these reasons, the hypotheses on which the research is based were formed as follows;

H11 hypothesis: The diabetic foot school program applied in diabetic foot patients has an effect on foot biomechanical measurements and gait parameters.

Hypothesis H12: In diabetic foot patients, the diabetic foot school program has an effect on the sensation of individuals.

H13 hypothesis: In diabetic foot patients, the diabetic foot school program has an effect on the balance of individuals.

H14 hypothesis: In diabetic foot patients, the diabetic foot school program has an effect on the diabetic foot and self-care behaviors of individuals.

DETAILED DESCRIPTION:
The study will be carried out in a special gait analysis center. To work; Volunteers, aged 40-70 years, diagnosed with diabetic foot and having type 2 diabetes mellitus with neuropathic symptoms will be included. Participants will be randomly divided into two groups before starting. Trainings will be given to the 1st group within the scope of diabetic foot school, and an exercise program aiming to increase the mobility and strength of the foot will be implemented through video calls twice a week, face-to-face once a week for 8 weeks. The 2nd group will be given a booklet covering this training and they will be followed up with video calls 1 day a week for 8 weeks. In diabetic foot school education, foot anatomy and functions, biomechanics, diabetic foot causes, epidemiology, causes of pain will be explained and treatment methods, ergonomic information, exercises to be done, sensory education, appropriate positions in daily life activities, risky situations, points to be considered and foot care. information will be given.

Before the research, individuals will be informed about the purpose and content of the study.

Ulcer advanced to Wagner grade 3,4 or 5, standardized mini mental state assessment scale score below 18 points, body mass index over 30, gestational diabetes, malignant tumor, neurological and exacerbated systemic disease, charcot neuroarthropathy, length difference in the lower extremity, fracture, surgical operation and Individuals who have received training on diabetic foot before and who have received other treatments that may affect wound healing will be excluded from the study.

All evaluations of both groups will be made by the same physiotherapist before and 8 weeks after the study. At the end of the study, individuals in the 2nd group will be included in the diabetic foot school training upon their wishes.

Within the scope of the study, information such as demographic information, smoking status, medical history, ulcer history, previous ulcer locations, if any, medications they use, walking aids/orthotics/diabetic shoes, existing foot deformities will be recorded and Plantar pressure senses; With Semmes-Weinstein monofilaments, Vibration sense; With 128 Hz tuning fork, Pain; with neuropathic pain questionnaire (DN4) and visual analog scale (VAS), lower extremity position sense (proprioception sense); Acumar dual digital inclinometer, Lower extremity muscle strengths (hip flexor, extensor, knee flexor, extensor and ankle plantar flexor and dorsi flexors) with HandHeld Dynamometer muscle dynamometer, Lower extremity strengths with 'Stair Climbing Test (MICT)', their balance; With the 'Get Up and Walk Test' and the 'Functional Reach Test', The time-distance characteristics of the gait will be evaluated by means of a motion-detecting wireless sensor, BTS-G (G Sensor, BTS Bioengineering S.p.A., Italy).

Plantar pressures during walking will be evaluated with Rsscan (v9 clinical 2mt plate advanced system) pedobarography.

Individuals' knowledge about diabetic foot will be evaluated face to face with diabetic foot knowledge scale, foot self-care behaviors, diabetic foot self-care questionnaire and foot care behavior scale.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetic foot between the ages of 40-70,
* Type 2 diabetes patients with neuropathic symptoms
* standard wound care protocol is applied (cleaning the wound with saline, covering it with gauze),
* sedentary who has not exercised regularly for six months,
* Able to walk at least 10 meters unaided,
* Volunteers

Exclusion Criteria:

* Ulcer that has progressed to Wagner grade 3,4 or 5,
* standardized mini mental state assessment scale score below 18 points,
* body mass index over 30,
* gestational diabetes mellitus,
* malignant tumor,
* neurological and exacerbated systemic disease,
* Charcot neuroarthropathy,
* length difference in lower extremity, fracture, surgical operation and
* Individuals with previous training in diabetic foot and other treatments that may affect wound healing

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Plantar pressure senses | immediately after the intervention.
  With Semmes-Weinstein monofilaments, In order to understand the test, individuals will be placed on the patient bed with their feet bare in the supine position, and several different points on the soles of the feet will be touched with a thick filament, first with the eyes open and then with the eyes closed, and the individual will be asked to answer "yes" when they feel the filament touch. . With each filament, each test point on the sole of the foot will be held for 2 seconds by applying pressure 3 times at right angles until the filament bends, and when the individual knows 1 of these 3 touches correctly, the relevant filament thickness will be recorded as the light touch-pressure threshold value for that test point of the individual.

SECONDARY OUTCOMES:
Vibration sense | immediately after the intervention
  It will be evaluated over the first metatarsal head and medial malleolus with a 128 Hz tuning fork. The test will be explained by positioning the individuals as in other tests, and the actual evaluations will begin after the individual expresses that he/she understands the test. The physiotherapist will sit on a chair at the foot of the patient and touch the fork to the test point in an upright position, immediately after hitting the tip of the tuning fork to the foot. In the meantime, the individual was asked to say "done" as soon as he did not feel the vibration by running the digital stopwatch. The stopwatch will be stopped when the individual says "done". Evaluation will be applied 3 times for each test point and the average of the time obtained from the three applications will be recorded as the individual's vibration sense score.

OTHER OUTCOMES:
Patient's Pain | immediately after the intervention
  will be evaluated with the neuropathic pain questionnaire (DN4). The DN-4 questionnaire was developed by the French Neuropathic Pain Group as a clinical-based questionnaire to describe pain with a neuropathic character. The DN-4 questionnaire consists of 10 items; While the first seven items are related to the patient's subjective sensory complaints, the last three items are related to clinical findings. Patients with a DN-4 score of ≥4 are considered to have neuropathic pain. DN4 contains 7 questions about symptoms and 3 questions about clinical treatment. The DN4 scoring is an easy tool and a total score of 4 out of 10 or above indicates neuropathic pain. The higher the score, the greater the pain. The questionnaire was validated for neuropathic pain screening in patients with painful diabetic neuropathy, and its Turkish validation was done by Ünal Çevik.
Patient's Pain | immediately after the intervention
  will be evaluated with the visual analog scale (VAS). VAS subjects will be asked to mark the pain they feel on a horizontal line between 0-100 mm, after explaining that 0 mm means "no pain" and 100 mm means "the most severe" pain. Then the marked distance will be measured from the left end with a ruler and recorded.
lower extremity position sense (proprioception sense); | immediately after the intervention
  will be evaluated with a dual digital inclinometer. During the test, measurements will be performed by placing the inclinometer parallel to the foot, with the individuals in the supine position, with their eyes closed to avoid visual cues. While determining the target angles, the angles that are frequently used in the studies in the literature and that are functional in walking will be preferred. Individuals will be told to focus on the position of the ankle joints in space for 5 seconds by bringing their feet in the neutral position to the target position, and by repeating this process 3 times, the patient will learn this position. Then, the individual was asked to repeat the target angle during the testing phase. Measurements will be repeated 3 times for each target angle. As a result criterion; recording the absolute value of the deviation amounts from the target angles; The average of the deviations occurring during the 3 repetitions will be taken.
Lower extremity muscle strengths | immediately after the intervention
  (hip flexor, extensor, knee flexor, extensor and ankle plantar flexor and dorsi flexors) will be evaluated with the HandHeld Dynamometer muscle dynamometer. Hand-held dynamometers are easy to use compared to isokinetic devices due to their simple, convenient portability, cost and small size, and are accepted as a reliable and valid tool for evaluating muscle strength in the clinical setting. During the test, the "make test" technique, which requires isometric contraction, will be applied. (Make test, while the measurer is holding the dynamometer steady, against the maximum force application protocol)
Lower extremity strengths | immediately after the intervention
  It will be evaluated with the 'Stair Climbing Test (MICT)'. In MICT, the patient will first be asked to climb 9 steps with a step height of approximately 20 cm, then return and descend 9 steps. If the patient used the assistive device during the test, it will be noted. The time the test is completed will be measured with a stopwatch and recorded in seconds.
balance | immediately after the intervention
  It will be evaluated with the 'Get Up and Go Test'. This test is a valid, reliable, practical method that does not require any special equipment to evaluate functional mobility. It measures the time required to complete some functional tasks and is also used in determining the risk of falling. The test is carried out at a distance of 3 meters. Individuals are asked to get up from the sitting position in the chair, walk a distance of 3 meters, come back and sit again, and the elapsed time is recorded.
balance | immediately after the intervention
  It will be evaluated with the 'Functional Reach Test'.It is a test that identifies the ability to reach with the upper extremity while maintaining trunk stability. It provides the evaluation of the balance in daily activities. For the evaluation, the individual will first be asked to extend his arm straight forward and the distance they have reached will be recorded, then they will be asked to reach forward as far as they can without getting their heels off the ground, and the maximum value they can reach without losing their balance will be marked. This measurement will be repeated three times and averaged.
The time-distance characteristics of the gait | immediately after the intervention
  will be evaluated by means of a motion-detecting wireless sensor, BTS-G (G Sensor, BTS Bioengineering S.p.A., Italy).
  The sensor, which is attached to the waist of the individuals with the help of a semi-elastic belt surrounding the lumbal 4-5 intervertebral spaces, transfers the acceleration data in the anteroposterior, mediolateral and vertical axes to the computer via bluetooth. The system compares the data from the right and left extremities with normal values during walking and also performs a kinematic analysis of the pelvis in 3 planes. In our study, individuals will be asked to walk as normally as possible at a pace of their own choosing, and data on the time-distance characteristic of their gait will be collected.
Plantar pressures during walking | immediately after the intervention
  will be evaluated with ('Rsscan v9' clinical 2mt plate advanced system) pedobarography. The data obtained with the device is: maximum pressure (N/cm2). Individuals will be asked to walk at normal walking speeds on a flat platform and foot and gait analyzes will be made through the computer program.
Individuals' information about diabetic foot | immediately after the intervention.
  Diabetic foot knowledge scale; Diabetic foot knowledge will be evaluated using the 5-item Diabetes Foot Care Knowledge Scale, which is a subscale of Diabetes Knowledge Qustionnaire-24. While calculating the DABÖ score, the correct and incorrectly coded yes answers are given a score of 1, and the other situations are given a score of 0. The closer the average score is to 5, the better the level of knowledge.
Individuals' information about diabetic foot | immediately after the intervention.
  was determined by diabetic foot self-care questionnaire. Diabetic foot self-care questionnaire; It is a likert type scale developed by Bonnie Elliott Quarles in 2005 in accordance with western culture to determine the perception of diabetic patients' self-perception of diabetic foot care activities. Self-efficacy is measured by scoring between 0 and 10. The scale consists of 9 items. The 9 statements that make up the scale are evaluated on the 11-digit visual scale, which is stated as -I'm not sure at all=0 and I'm very sure=10. The lowest score of the scale is 0, and the highest score is 100.
Individuals' information about diabetic foot | immediately after the intervention.
  was determined by diabetic foot self-care questionnaire and foot care behavior scale. The Foot Care Behavior Scale was created by Borges in 2007 with 16 items in line with the criteria of the American Diabetes Association (ADA) in order to develop foot self-care behaviors. In the study, the language validity of the observation guide was made into Turkish and it was adapted as a 15-item Foot Care Behavior Scale in line with expert opinions. In each interview with the patients, their foot care behaviors were evaluated in line with this guideline. The rating is (1=Never, 2=Sometimes, 3=Sometimes, 4=Often, 5=Always)

CONTACTS AND LOCATIONS:
Overall Officials: Bahar KÜLÜNKOĞLU, assc. prof., Study Director — Ankara Yildirim Beyazıt University

IPD SHARING:
Plan to Share IPD: No